CLINICAL TRIAL: NCT00347334
Title: Is Home Positioning Time Associated With Torticollis Rate of Recovery?
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Other Study IDs: 05-209
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Torticollis
Keywords: Torticollis; infant home positioning; head control
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: infant home positioning

SUMMARY:
The term torticollis is Latin for "twisted neck". It can be caused by a tightness of the sternocleidomastoid muscle manifested by a head tilt to the same and neck rotation to the opposite side. Treatment includes a comprehensive physical therapy program. Torticollis typically presents itself within the first three months of life. Currently research in infants concludes that a physical therapy stretching program is effective in the majority of cases.1

The study will determine how positioning time correlates to rate of recovery. Overall incidence of torticollis has increased dramatically since the inception of the back to sleep program in 1994.2 The back to sleep program is an educational awareness program promoting families to place infants to sleep on their backs to reduce the risks of sudden infant death. The increase use of semi-upright positioning equipment prior to developmental head control may also be contributing to the increase. Families are placing babies in semi-upright position ie. car seat or swing prior to developmental head control. Head control typically emerges by three months of age. Unfortunately the use of positioning devices occurs prior to the child reaching their third month birthday.

The specific aims of the study will include measuring the rate of recovery for infant torticollis. Recovery will be defined as achieving full neck rotation and no head tilt. The length of time spent in developmental positions and positioning equipment such as belly lying, side lying, semi-upright and sitting will also be monitored and recorded. No specific position will be prescribed; the study will monitor positions only.

Treatment will be initiated upon referral to Cleveland Clinic Children's Hospital for physical therapy evaluation. Baseline for cervical rotation and lateral tilt will be assessed. Families will be trained regarding a home stretching program and asked to diary home positioning time. Routine plan of care will continue a minimum of every other week until full active range of motion is achieved. At each visit cervical range of motion will be determined as well as parent report regarding home positioning time. Recovery will be defined as full active range of motion, no head tilt, and symmetrical head righting reactions. Post recovery analysis of recovery rates and positioning time will be done to assess correlations.

DETAILED DESCRIPTION:
Torticollis come from Latin,"torti" meaning twisted and "collis" meaning neck.1 Torticollis is a tightening of sternocleidomastoid (SCM) muscle resulting in a head tilt to involved side and rotation to the opposite side. The conditions presents from birth through the first 2 months of life during which time infants' neck muscles are developing. There are three clinical groups of torticollis-

1. palpable SCM tumor
2. muscular SCM- tightening and thickening of SCM
3. postural torticollis - posturing but no tightness or tumor 2 The causes of torticollis may include damage or shortening of SCM possibly due to: in utero positioning ie. lack of space traumatic birth multiple birth therefore limiting space low amniotic fluid

Current physical therapy referrals for torticollis have increased dramatically perhaps due to an increase in multiple births, infant size and premature birth. Graham states that the back to sleep program initiated in 1994 has resulted in an epidemic of plagiocephaly and positional torticollis estimated from 1 in 300 to 1 in 60.3 In addition the increase use of infant seats places children in semi-upright postures before an age of developmental head control.

Current research has established that physical therapy is effective in 90% of the cases. The treatment is correlated with severity of restriction and the presence of tumor.4 The role of home positioning has not been addressed in torticollis research. A community education program to promote awareness limiting time in a semi-upright position ie. could help decrease the surge of torticollis.

The study significance is to establish how home positioning time correlates to rate of recovery for Torticollis. Does positioning the child out of semi-upright improve recovery rates? Can we establish a better physical therapy intervention? This improves quality of physical therapy care.

Specific Aims:

At this point physical therapy research interventions for Torticollis have focused on a stretching program. This study will determine how home positioning correlates to the torticollis rate of recovery. The hypothesis is to determine the relationship between developmental positions and rate of recovery for Torticollis. Does home positioning affect recovery? Recovery will be determined by time to achieve full active range of motion and symmetrical head control as measured by a goniometer.

The aims include measuring Torticollis recovery time, documenting neck movements using a goniometer, a standardized physical therapy measurement tool. As well as recording home positioning through parent report. All participants will be consented prior to treatment.

Experimental Design and Methods:

A prospective observational design study to determine: Is home positioning time associated with torticollis rate of recovery? Infants with a torticollis diagnosis, six months of age or younger, referred to Cleveland Clinic Children's Hospital will be eligible for the study to obtain a sample of 150 children. A marketing campaign to locale physicians will educate them regarding the study existence at the four satellite locations. The study will explore the relationship between home positioning times and recovery rates.

Infants will be followed a minimum of every other week to assess active and passive neck and trunk range of motion, head and neck control including strength and righting reactions. Parents will diary reporting weekly time spent in developmental postures: back, side belly, and semi-upright posture ie. infant car seat. Postures will advance with developmental age to sitting.

Physical therapy interventions during weekly sessions include routine plan of care:

stretching of neck and trunk strengthening of neck and trunk kineseotaping of neck and trunk Parent education regarding home stretching and environmental adaptation Massage/Soft tissue mobilization and myofascial release to head and trunk Environmental adaptation encourage child to look the opposite Orthotic management - Tot collar use

Protocols for taping and stretching will be followed. A tubular orthosis for Torticollis (TOT collar) will be utilized at 4.5 months if a head tilt is still present at this age.

Once full passive range of motion is achieved treatment will progress to address active range of motion, strengthening as well as postural asymmetries.

A standardized torticollis assessment, plan of care and weekly note will be used by all clinicians for documentation. Staff training will occur prior to initiation of study and quarterly throughout the study. These training will be videotaped and all clinicians will be required to view prior to treatment.

Plagiocephaly often accompanies infants with torticollis. Referral to craniofacial physician for helmeting consultation will occur at 6 months of age if indicated. Plagiocephaly is a flattened head due to asymmetrical resting posture of the infant. Plagiocephaly will be defined as greater than a 4mm cross sectional difference.

Recovery is defined as :

1. Full symmetrical active range of motion of neck, trunk and extremities as measured by goniometry per Norkin.5
2. 80* active cervical rotation in supine, prone, sitting and stance as measured by goniometry.
3. Active midline trunk and head alignment during static and dynamic activity
4. Symmetrical righting and equilibrium reactions.
5. Symmetrical antigravity head and trunk strength as measured by manual muscle strength testing by Hoppenfeld.6

Data:

The primary outcome variables are rate of recovery as defined by length of time from recovery and initial assessment. Positioning time spent in developmental postures: belly, back, semi-upright and sit. Other parameters which will be documented are: age of parents, birth weight, birth order, multiple births: yes or no, plagiocephaly, helmet use and TOT collar use. Data will be coded and recorded on an Excel spreadsheet. Reports will be recorded aggregately.

Statistical methods:

We will assess the relationship between recovery time and positioning time in each position using Pearson's correlation coefficient or the non-parametric Spearman rank correlation coefficient as necessary. We will use multiple linear regression models to assess these relationships while adjusting for baseline and treatment factors such as birth order, plagiocephaly and TOT collar use. All tests will be two-tailed and performed at a significance level of 0.05. All analyses will be performed using SAS 9.1 software (SAS institute, Cary NC)

Sample Size: With the 150 subjects we anticipate, we will have greater than 90% power to detect correlation coefficient of at least 0.30.

Inclusion/Exclusion:

A full medical assessment is necessary to rule out associated anomalies such as hip dysplasia, vertebral anomalies due to syndromes ie. Down's syndrome. A secondary diagnosis often associated with torticollis is plagiocephaly. Asymetrical resting posture often results in a flattened head (plagiocephaly). This may cause a progressive cranial asymmetry. In some cases plagiocephaly requires helmeting to apply pressures and reshape the infants head. Children with vertebral anomalies will be excluded; children will plagiocephaly will be included.

Treatment for torticollis primarily includes physical therapy interventions. Ninety percent of cases respond to physical therapy. In severe cases when after a six month stretching program there still remains greater than 15* head tilt more aggressive treatment may be indicated. Other interventions include Botulinum Toxin injection to weaken the muscle and possibly surgery to lengthen the muscle.4

Exclusion criteria include:

treatment initiated at another facility medical complication interfered with treatment surgery radiology results of vertebral anomaly, ocular imbalance or nerve injury treatment initiated after six months of age previous BOTOX or cervical manipulations clients who attend daycare full time compliance with less than 80% scheduled sessions.

Study procedures:

Participants will receive routine plan of care. Additional procedures required for participants include completing a diary/questionnaire regarding home positioning.

Consent

Consent will be attained by treating physical therapist prior to initial assessment.

1. Powell,F. The effects of kinesio taping method in treatment of congenital torticollis case studies. 62-75.
2. Cheng JC, Wong MW, Tand SP, Chen TM, Shum SL, Wong EM. Clinical determinants of the outcome for manual stretching in the treatment of congenital torticollis in infants. J bone Joint Surg AM. 2001 May:83-A: 679-87.
3. Graham JM Management of Plagiocephaly and Torticollis CSMS Pediatrics/Medical Genetics 3/14/01.
4. Emery C. The determinants of treatment duration for congenital muscular torticollis. Phys Ther. 1994 Oct:74(10):921-9.
5. Norkin CC, White DJ, Measurement of joint motion: a guide to goniometry. FA Davis Co. 1985
6. Hoppenfeld S, Physical Examination of the Spine and Extremities. Appleton-Century-Crofts, 1976.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of torticollis
* 6 months of age or less

Exclusion Criteria:

* previous surgery
* treatment initiated at another facility
* medical complication which interfere with treatment
* radiology results of vertebral anomaly, ocular imbalance of nerve injury
* compliance with less than 80% scheduled sessions

Ages: 5 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie S Pace, MPT, Principal Investigator — Cleveland Clinic Foundation - Children's Hospital
Locations (3):
- United States (3):
  - Cleveland Clinic Children's Hospital - East location, Beachwood, Ohio
  - Cleveland Clinic Children's Hospital - Shaker campus, Cleveland, Ohio
  - Cleveland Clinic Children's Hospital - Westlake, Westlake, Ohio